CLINICAL TRIAL: NCT02664792
Title: Use of [18]F-FDG - PET/CT in Brazil Unified Health System (SUS) as an Alternative Non-invasive Method for Staging of Lung Cancer
Brief Title: Use of [18]F-FDG on PET/CT as an Alternative Non-invasive Method for Staging of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Instituto do Cérebro do Rio Grande do Sul - InsCer (Unknown); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LACOG 0114
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Non-small Cell Lung Carcinoma
Keywords: Non-small cell lung carcinoma; PET/CT; 18F-FDG
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnosis or suspicion of non-small cell lung carcinoma (Experimental): SUS patients with diagnosis or suspicion of non-small cell lung carcinoma with an indication for mediastinoscopy
  Interventions: Other: Use of [18f]FDG - PET/CT for the diagnosis and staging of non-small cell lung carcinoma

INTERVENTIONS:
Other: Use of [18f]FDG - PET/CT for the diagnosis and staging of non-small cell lung carcinoma

SUMMARY:
To evaluate the diagnostic accuracy of the 18Fluor-fluorodeoxyglucose ([18F]FDG) in the Positron Emission Tomography/Computed Tomography (PET/CT) as compared to mediastinoscopy for staging of non-small cel lung carcinoma.

DETAILED DESCRIPTION:
The main aim of this study is to validate the [18F]FDG on PET/CT for the diagnosis of metastatic ganglions at the mediastinum in SUS patients with non-small cell lung carcinoma considering sensitivity, specificity, positive predictive value, negative predictive value, accuracy. Other specific aims are:

* Analyze the diagnosis performance of the [18F]FDG on PET/CT in two timepoints (1 and 2 hours after exam), in relation to the staging of the non-small cell lung carcinoma
* Evaluate the addition of the iodinated contrast in the [18F]FDG to improve the images obtained from the PET/CT in the staging of the non-small cell lung carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with histological diagnosis or high suspicion of non-small cell lung carcinoma
2. Patients who previously underwent staging of the disease with CT
3. Clinical stages I-III AJCC 7th edition.
4. Patients with indication for mediastinoscopy and linfonodal biopsy
5. Patients without treatment for lung cancer
6. Patients with biochemical and haematological exams
7. Women of childbearing potential using contraceptive methods and negative pregnancy test
8. Adults with more than 18 years old.
9. Both genders

Exclusion Criteria:

* Pregnant women
* Patients with other types of patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Validate the [18F]FDG as an alternative method for non-small lung carcinoma diagnosis | 4 years

SECONDARY OUTCOMES:
Number of patients diagnosed in a positive manner with the gold standard and with the alternative method | up to 30 days following recruitment
Number of patients with a negative diagnosis according to the gold standard and the alternative method | up to 30 days following recruitment
Number of true positives among positive diagnosed patients with the alternative method | up to 30 days following recruitment
Number of false positives among patients negatively diagnosed with the alternative method | up to 30 days following recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Werutsky, MD, Study Director — Latin American Cooperative Oncology Group
Locations (1):
- Instituto do Cérebro do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alberg AJ, Ford JG, Samet JM; American College of Chest Physicians. Epidemiology of lung cancer: ACCP evidence-based clinical practice guidelines (2nd edition). Chest. 2007 Sep;132(3 Suppl):29S-55S. doi: 10.1378/chest.07-1347. PMID 17873159
- [Background] Alberg AJ, Samet JM. Epidemiology of lung cancer. Chest. 2003 Jan;123(1 Suppl):21S-49S. doi: 10.1378/chest.123.1_suppl.21s. PMID 12527563
- [Background] Molina JR, Yang P, Cassivi SD, Schild SE, Adjei AA. Non-small cell lung cancer: epidemiology, risk factors, treatment, and survivorship. Mayo Clin Proc. 2008 May;83(5):584-94. doi: 10.4065/83.5.584. PMID 18452692
- [Background] Nana-Sinkam SP, Powell CA. Molecular biology of lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e30S-e39S. doi: 10.1378/chest.12-2346. PMID 23649444
- [Background] Daigo Y, Takano A, Teramoto K, Chung S, Nakamura Y. A systematic approach to the development of novel therapeutics for lung cancer using genomic analyses. Clin Pharmacol Ther. 2013 Aug;94(2):218-23. doi: 10.1038/clpt.2013.90. Epub 2013 May 8. PMID 23657161
- [Background] Sommer G, Wiese M, Winter L, Lenz C, Klarhofer M, Forrer F, Lardinois D, Bremerich J. Preoperative staging of non-small-cell lung cancer: comparison of whole-body diffusion-weighted magnetic resonance imaging and 18F-fluorodeoxyglucose-positron emission tomography/computed tomography. Eur Radiol. 2012 Dec;22(12):2859-67. doi: 10.1007/s00330-012-2542-y. Epub 2012 Jul 9. PMID 22772365
- [Background] Miller PW, Long NJ, Vilar R, Gee AD. Synthesis of 11C, 18F, 15O, and 13N radiolabels for positron emission tomography. Angew Chem Int Ed Engl. 2008;47(47):8998-9033. doi: 10.1002/anie.200800222. PMID 18988199
- [Background] Leitha T. Nuclear medicine: proof of principle for targeted drugs in diagnosis and therapy. Curr Pharm Des. 2009;15(2):173-87. doi: 10.2174/138161209787002898. PMID 19149611
- [Background] Fowler JS, Ido T. Initial and subsequent approach for the synthesis of 18FDG. Semin Nucl Med. 2002 Jan;32(1):6-12. doi: 10.1053/snuc.2002.29270. PMID 11839070
- [Background] Zanzonico P. Basic Sciences of Nuclear Medicine. Med Phys. 2011 Sep;38(9):5265-5266. doi: 10.1118/1.3626488. No abstract available. PMID 28524975
- [Background] March 10, 2000 Federal Register, Docket No 00N-0553, p.p. 12999-13010
- [Background] VALLABHAJOSULA, S. Molecular Imaging: radiopharmaceuticals for PET and SPECT. New York: Springer, 2009. 371p.
- [Background] Murray CJ, Atkinson C, Bhalla K, Birbeck G, Burstein R, Chou D, Dellavalle R, Danaei G, Ezzati M, Fahimi A, Flaxman D, Foreman, Gabriel S, Gakidou E, Kassebaum N, Khatibzadeh S, Lim S, Lipshultz SE, London S, Lopez, MacIntyre MF, Mokdad AH, Moran A, Moran AE, Mozaffarian D, Murphy T, Naghavi M, Pope C, Roberts T, Salomon J, Schwebel DC, Shahraz S, Sleet DA, Murray, Abraham J, Ali MK, Atkinson C, Bartels DH, Bhalla K, Birbeck G, Burstein R, Chen H, Criqui MH, Dahodwala, Jarlais, Ding EL, Dorsey ER, Ebel BE, Ezzati M, Fahami, Flaxman S, Flaxman AD, Gonzalez-Medina D, Grant B, Hagan H, Hoffman H, Kassebaum N, Khatibzadeh S, Leasher JL, Lin J, Lipshultz SE, Lozano R, Lu Y, Mallinger L, McDermott MM, Micha R, Miller TR, Mokdad AA, Mokdad AH, Mozaffarian D, Naghavi M, Narayan KM, Omer SB, Pelizzari PM, Phillips D, Ranganathan D, Rivara FP, Roberts T, Sampson U, Sanman E, Sapkota A, Schwebel DC, Sharaz S, Shivakoti R, Singh GM, Singh D, Tavakkoli M, Towbin JA, Wilkinson JD, Zabetian A, Murray, Abraham J, Ali MK, Alvardo M, Atkinson C, Baddour LM, Benjamin EJ, Bhalla K, Birbeck G, Bolliger I, Burstein R, Carnahan E, Chou D, Chugh SS, Cohen A, Colson KE, Cooper LT, Couser W, Criqui MH, Dabhadkar KC, Dellavalle RP, Jarlais, Dicker D, Dorsey ER, Duber H, Ebel BE, Engell RE, Ezzati M, Felson DT, Finucane MM, Flaxman S, Flaxman AD, Fleming T, Foreman, Forouzanfar MH, Freedman G, Freeman MK, Gakidou E, Gillum RF, Gonzalez-Medina D, Gosselin R, Gutierrez HR, Hagan H, Havmoeller R, Hoffman H, Jacobsen KH, James SL, Jasrasaria R, Jayarman S, Johns N, Kassebaum N, Khatibzadeh S, Lan Q, Leasher JL, Lim S, Lipshultz SE, London S, Lopez, Lozano R, Lu Y, Mallinger L, Meltzer M, Mensah GA, Michaud C, Miller TR, Mock C, Moffitt TE, Mokdad AA, Mokdad AH, Moran A, Naghavi M, Narayan KM, Nelson RG, Olives C, Omer SB, Ortblad K, Ostro B, Pelizzari PM, Phillips D, Raju M, Razavi H, Ritz B, Roberts T, Sacco RL, Salomon J, Sampson U, Schwebel DC, Shahraz S, Shibuya K, Silberberg D, Singh JA, Steenland K, Taylor JA, Thurston GD, Vavilala MS, Vos T, Wagner GR, Weinstock MA, Weisskopf MG, Wulf S, Murray; U.S. Burden of Disease Collaborators. The state of US health, 1990-2010: burden of diseases, injuries, and risk factors. JAMA. 2013 Aug 14;310(6):591-608. doi: 10.1001/jama.2013.13805. PMID 23842577
- [Background] Gould MK, Kuschner WG, Rydzak CE, Maclean CC, Demas AN, Shigemitsu H, Chan JK, Owens DK. Test performance of positron emission tomography and computed tomography for mediastinal staging in patients with non-small-cell lung cancer: a meta-analysis. Ann Intern Med. 2003 Dec 2;139(11):879-92. doi: 10.7326/0003-4819-139-11-200311180-00013. PMID 14644890
- [Background] Bille A, Pelosi E, Skanjeti A, Arena V, Errico L, Borasio P, Mancini M, Ardissone F. Preoperative intrathoracic lymph node staging in patients with non-small-cell lung cancer: accuracy of integrated positron emission tomography and computed tomography. Eur J Cardiothorac Surg. 2009 Sep;36(3):440-5. doi: 10.1016/j.ejcts.2009.04.003. Epub 2009 May 22. PMID 19464906
- [Background] Product Information: Fludeoxyglucose F18 IV injection, Fludeoxyglucose F18 IV injection. Feinstein Institute for Medical Research, Manhasset, NY, 2010.
- [Background] Jones SR, Carley S, Harrison M. An introduction to power and sample size estimation. Emerg Med J. 2003 Sep;20(5):453-8. doi: 10.1136/emj.20.5.453. PMID 12954688
- [Background] Erasmus JJ, McAdams HP, Patz EF Jr, Goodman PC, Coleman RE. Thoracic FDG PET: state of the art. Radiographics. 1998 Jan-Feb;18(1):5-20. doi: 10.1148/radiographics.18.1.9460106.
- [Background] Singh J, Daftary A. Iodinated contrast media and their adverse reactions. J Nucl Med Technol. 2008 Jun;36(2):69-74; quiz 76-7. doi: 10.2967/jnmt.107.047621. Epub 2008 May 15. PMID 18483141
- [Derived] Werutsky G, Hochhegger B, Lopes de Figueiredo Pinto JA, Martinez-Mesa J, Zanini ML, Berdichevski EH, Vilas E, da Silva VD, Tsukazan MTR, Vieira A, Fritscher LG, Hartmann L, Alba M, Sartori G, Matushita C, Bortolotto V, do Amaral RR, Junior LCA, Zaffaroni F, Barrios CH, Debiasi M, Frietscher CC. PET-CT has low specificity for mediastinal staging of non-small-cell lung cancer in an endemic area for tuberculosis: a diagnostic test study (LACOG 0114). BMC Cancer. 2019 Jan 3;19(1):5. doi: 10.1186/s12885-018-5233-5. PMID 30606144